CLINICAL TRIAL: NCT06079008
Title: The Association of Cardiac Valve Calcification and 1-year Mortality After Lower-extremity Amputation in Diabetic Patients: a Retrospective Study
Brief Title: The Association of Cardiac Valve Calcification and 1-year Mortality After Lower-extremity Amputation in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-035-01
Record Dates: First submitted 2023-05-17; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-01

CONDITIONS: Amputation; Diabetic Foot; Valve Disease, Aortic; Valve Heart Disease
MeSH Terms: conditions — Diabetic Foot; Aortic Valve Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survival group: The patients who survived more than 1-year after amputation surgery.
  Interventions: Other: calcified cardiac valve
- mortality group: The patients who were dead within 1-year after amputation surgery.
  Interventions: Other: calcified cardiac valve

INTERVENTIONS:
Other: calcified cardiac valve — patients have cardiac cardiac valve before surgery

SUMMARY:
The goal of this observational study is to learn about the association between cardiac valve calcification and the 1-year mortality after lower-extremity amputation in diabetic patients. Diabetic patients requiring lower-extremity amputation were retrospectively studied. Preoperative detailed anamnesis was taken. Cardiac valve calcification was assessed using echocardiography at baseline. One-year follow-up was conducted and included clinical visits, hospital record assessment, and telephone reviews to obtain the survival status of patients. Researchers compare the survival group to the mortality group to study the relationship between the cardiac valve calcification and mortality.

DETAILED DESCRIPTION:
This study aimed to investigate the association between cardiac valve calcification and 1-year mortality in diabetic patients after lower-extremity amputation. The investigator recruited consecutive patients who were admitted to the Sun Yat-sen Memorial Hospital for diabetic foot ulcers that needed amputation surgery. Clinical characteristics of each patient and the laboratory examination were collected before surgery. Cardiac valve calcification was assessed at baseline. This study obtained the survival status of patients within one year through outpatient follow-up and telephone follow-up. Researchers compared the survival group to the mortality group to see if the mortality group had a higher prevalence of heart valve calcification.

ELIGIBILITY:
Inclusion Criteria:

* Had echocardiography at baseline
* With diabetic foot ulcers that required amputation after orthopedist's assessment

Exclusion Criteria:

* Fractures due to traumatic reasons that required extremity amputation
* Amputation level below the ankle
* Severe sepsis that required vasoactive agent treatment
* Rheumatic heart disease
* Heart valve surgery history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator recruited consecutive patients who were admitted to the Sun Yat-sen Memorial Hospital for diabetic foot ulcers that needed amputation surgery between July 2017 and March 2021 and were followed up for 1 year after amputation surgery
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The proportion of cardiac valve calcification between survival group and mortality group | 2017-12-1
  The prevalence of calcified heart valve diseases was compared between the mortality group and survival group.

IPD SHARING:
Plan to Share IPD: No